CLINICAL TRIAL: NCT03824327
Title: A Phase I Trial Combining Papaverine and Stereotactic Body Radiation Therapy for Non-Small Cell Lung Cancer or Lung Metastases
Brief Title: Papaverine and Stereotactic Body Radiotherapy (SBRT) for Non Small Cell Lung Cancer (NSCLC) or Lung Metastases
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Jeremy Brownstein, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-18215; NCI-2019-00105 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-01-23; First posted 2019-01-31 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Papaverine; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (BOLD fMRI, papaverine hydrochloride, SBRT) (Experimental): Patients undergo BOLD fMRI and receive papaverine hydrochloride IV on days -7 to day 1. Within 30-90 minutes, patients undergo a second BOLD fMRI. Patients then receive papaverine hydrochloride IV and within 30-90 minutes after dose undergo SBRT for a up to 4-5 sessions over 2 weeks. Patients undergo CT scan throughout the study and blood sample collection on study.
  Interventions: Procedure: Blood Oxygen Level Dependent Imaging; Drug: Papaverine Hydrochloride; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Procedure: Blood Oxygen Level Dependent Imaging — Undergo BOLD fMRI
  Other Names: Blood Oxygen Level Dependent Functional Magnetic Resonance Imaging; BOLD; BOLD fMRI
Drug: Papaverine Hydrochloride — Given IV
  Other Names: Cerebid; Cerespan; Pap H; Pavabid; Pavacap; Therapav; Vasal; Vaso-Pav; Vasospan
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase I trial studies the side effects and how well papaverine hydrochloride and stereotactic radiation therapy body (SBRT) work in treating patients with non-small cell lung cancer. Papaverine hydrochloride may help radiation therapy work better by making tumor cells more sensitive to the radiation therapy. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Giving papaverine hydrochloride with SBRT may work in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of concurrent papaverine hydrochloride (PPV), and lung SBRT in patients with non-small cell lung cancer (NSCLC) or lung metastases.

SECONDARY OBJECTIVES:

I. To assess primary tumor control rate, local control rate, local-regional recurrence free-survival (LRRFS), disease-free survival (DFS), distant-metastasis-free survival (DMFS), and overall survival (OS).

II. To assess whether blood oxygen level-dependent (BOLD) functional magnetic resonance imaging (MRI) studies can predict which patients may respond best to PPV + SBRT, and detect changes in oxygenation before and after PPV administration.

III. To assess whether blood-based micro ribonucleic acid (miRNA) biomarkers can predict which patients may respond best to PPV + SBRT.

OUTLINE: This is a dose-escalation study of papaverine hydrochloride.

Patients undergo BOLD functional magnetic resonance imaging (fMRI) and receive papaverine hydrochloride intravenously (IV) on day 1. Within 30-90 minutes, patients undergo a second BOLD fMRI. Patients then receive papaverine hydrochloride IV and within 30-90 minutes after dose undergo SBRT for a up to 4-5 sessions over 2 weeks.

After completion of study treatment, patients are followed up at 4-6 weeks, 3 and 6 months, 1 and 2 years, then every 3 months for 2 years, and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven NSCLC for whom SBRT to a single lesion has been chosen as the primary treatment modality (planned dose 50 Gy in 4-5 daily fractions). Patients with lung metastases from solid tumors are eligible.
* Patients must have a tumor =< 5 cm as defined by computed tomography (CT) largest axial dimension. Presence of adjacent nodules considered neoplastic in the same lobe or other ipsilateral lobe are allowed as long as the nodule(s) can be encompassed in an SBRT gross tumor volume (GTV) of =< 5 cm, within 1 isocenter. Multiple isocenters are not allowed
* No prior radiation resulting in overlapping fields
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Must be able to undergo correlative research MRIs
* No active connective tissue disease (scleroderma) or idiopathic pulmonary fibrosis (IPF)
* No history of complete atrioventricular block, hepatic dysfunction (e.g. cirrhosis), or priapism
* Within 30 days of registration: patients must have vital signs, history/physical examination, and laboratory studies (liver function tests, creatinine or creatinine clearance assessment)
* Life expectancy of at least 12 weeks in the opinion of investigator
* Women of child-bearing potential (WOCBP) must have a negative pregnancy test within 14 days of registration. Urine human chorionic gonadotropin (HCG) is an acceptable pregnancy assessment. Nursing women may participate only if nursing is discontinued, due to the possibility of harm to nursing infants from the treatment regimen
* Within 90 days of registration: pulmonary function tests (PFTs) including forced expiratory volume in 1 second (FEV-1) and diffusion capacity of the lung for carbon monoxide (DLCO)
* Albumin >= 2.5 g/dL (within 30 days of study registration)
* Total bilirubin =< 1.5 x upper limit of normal (ULN) (within 30 days of study registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN (within 30 days of study registration)
* Creatinine =< 1.5 x ULN or calculated creatinine >= 50 mL/min, calculated by the Cockcroft-Gault formula or 24-hour urine creatinine clearance >= 50 mL/min (within 30 days of study registration)

Exclusion Criteria:

* History of another malignancy

  * Exception: Subjects who have been disease-free for >= 3 years, or subjects with a history of localized prostate cancer, in situ carcinoma (e.g. breast, cervix, oral cavity), differentiated thyroid neoplasm, completely resected non-melanoma skin cancer, are eligible
* Any serious and/or unstable pre-existing medical disorder (aside from malignancy exception above), psychiatric disorder, or other conditions that could interfere with subject?s safety, obtaining informed consent or compliance to the study procedures, in the opinion of the investigator
* Pregnancy or breastfeeding: Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, the duration of study participation and for 4 months after the last dose of study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. No breastfeeding while patient is on study
* Patients with history of pneumonectomy
* Prior cytotoxic chemotherapy, molecularly-targeted agents (e.g. erlotinib, crizotinib), or immunotherapy unless >= 2 weeks from last dose. Patients can start chemotherapy, immunotherapy, or other systemic therapy after completion of SBRT, but this should be planned for ≥ 2 weeks from last SBRT dose.
* History of active connective tissue disease (scleroderma), idiopathic pulmonary fibrosis, pneumonitis
* Hepatic insufficiency resulting in jaundice and/or coagulation defects, or not meeting laboratory values (albumin, total bilirubin, AST/ALT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) | Up to 2 weeks
  Will employ the Bayesian optimal interval (BOIN) design to find the MTD.

SECONDARY OUTCOMES:
Primary tumor control | At 12 and 24 months after stereotactic body radiation therapy (SBRT) completion
  Primary tumor control is defined as the absence of primary tumor failure. Will be calculated and 95% exact binomial confidence interval will be provided.
Local control rate (primary tumor control + involved lobar control) | Up to 12 months after SBRT completion
  Local control is defined as the absence of local failure. Will be calculated and 95% exact binomial confidence interval will be provided.
Local-regional recurrence free-survival | From time of entry onto study until the time of documented local-regional recurrence or death, assessed up to 12 months after SBRT completion
  Will be summarized using Kaplan-Meier method.
Distant metastasis-free survival | Time from entry onto study until the time of documented metastatic recurrence or death, assessed up to 12 months after SBRT treatment
  Will be summarized using Kaplan-Meier method.
Disease-free survival | Time from entry onto study until the time of any documented disease recurrence or death, assessed up to 12 months after SBRT completion
  Will be summarized using Kaplan-Meier method.
Overall survival | Time from study entry until time of death from any cause, assessed up to 12 months after SBRT completion
  Will be summarized using Kaplan-Meier method.
Changes in magnetic resonance imaging (MRI) blood oxygen level-dependent (BOLD) response | Up to 4 hours
  Will be measured before and after papaverine hydrochloride (PPV) delivery by the percentage change in relaxation rate on MRI. Will also analyze biomarkers descriptively and graphically to assess trends in changes in these markers over time and the association with response. Exploratory comparisons of groups of patients based on response will involve the use of analysis of variance (ANOVA) for continuous data and categorical methods such as Fisher?s exact and chi-square tests for discrete data.
Change in hypoxia-inducible micro ribonucleic acids (miRNAs) | Up to 3 months
  Will analyze patient serum pre-and post-treatment for hypoxia-associated at pre- and post- SBRT treatment hypoxia-inducible microRNAs (miRs) using nanoString miRNA assay that could indicate the presence of tumor hypoxia. The changes in circulating biomarkers will be validated by alternative quantitative polymerase chain reaction (qPCR) based approaches. These results will be cross-validated with the BOLD data. Will also analyze biomarkers descriptively and graphically to assess trends in changes in these markers over time and the association with response. Exploratory comparisons of groups of patients based on response will involve the use of ANOVA for continuous data and categorical methods such as Fisher?s exact and chi-square tests for discrete data.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Brownstein, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu